CLINICAL TRIAL: NCT00480675
Title: Randomized Study Comparing Fluoroscopically-Guided Versus Blinded Trochanteric Bursa Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Johns Hopkins Office of Research Administration, Amanda Gibson
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00006986
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Bursitis
Keywords: bursitis; injection; fluoroscopy
MeSH Terms: conditions — Bursitis | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Trochanteric bursa injections done into the bursa under fluoroscopic guidance
  Interventions: Procedure: trochanteric bursa injection done under fluoroscopy with depomedrol and bupivacaine
- 2 (Active Comparator): Trochanteric bursa injection done with sham fluoroscopy using only landmarks as guidance.
  Interventions: Procedure: Trochanteric bursa injection with depomedrol and bupivacaine

INTERVENTIONS:
Procedure: trochanteric bursa injection done under fluoroscopy with depomedrol and bupivacaine — Depomedrol 60 mg + bupivacaine 2.5 ml
  Arms: 1
Procedure: Trochanteric bursa injection with depomedrol and bupivacaine — Trochanteric bursa injection done with sham x-ray and 60 mg of depomedroal and 2.5 ml bupivacaine using landmarks for guidance.
  Arms: 2

SUMMARY:
The goals of our research project are to study the relationship, if any, between the success of a TB injection (measured by pain relief and general patient satisfaction) and the method in which it was placed. Because fluoroscopy places patients requires a slight risk from radiation exposure and increased cost versus blind injection, it is important to know if there is an advantage to using this technique. The investigators will randomize 64 patients to receive either trochanteric bursa injections with corticosteroid and local anesthetic guided by fluoroscopy, or trochanteric bursa patients to receive trochanteric bursa injections based on landmarks on palpation. The investigators will then determine which method is superior, and whether injecting steroid and local anesthetic into the bursa itself is superior or inferior to injecting it into a tender area outside the bursa.

DETAILED DESCRIPTION:
This will be a randomized, controlled study evaluating the value of fluoroscopy in trochanteric bursa injections. Subjects will be recruited solely from the patients we normally see at the Blaustein Pain Treatment Center with a clinical diagnosis of GTPS. Sixty-four patients will be randomized in a 1:1 ratio using sealed envelopes to receive either TB corticosteroid injection done blind or with fluoroscopy. All patients who provide informed consent will be brought into the fluoroscopy suite and placed in the lateral decubitus position. In the patients randomized to receive fluoroscopically guided injections, a 22-gauge needle will be placed into the TB and correct position confirmed by fluoroscopy and contrast injection (1 ml per attempt) before corticosteroid and local anesthetic injection (60 mg of depomedrol and 2.5 ml of 0.5% bupivacaine). In the blinded group, one sham, pulsed fluoroscopic image will be taken of the femur, and the injection will be done based only on physical exam (overlying the area of maximal tenderness) and landmarks. Prior to the injection, 1 ml of contrast will be administered and another image taken to determine whether or not the needle is within the bursa, but this will not alter the injection. After contrast administration, the same corticosteroid and bupivacaine injection will be administered. The 2 main questions we propose to answer are: 1) whether using fluoroscopy for TB injections results in improved outcomes (comparison of the 32 patients in each group); and 2) whether injecting into the bursa provides superior results than performing non-bursal injections into the area of maximal tenderness (comparison of 32 patients who receive fluoroscopically-guided bursa injections + those patients whose blinded injection was noted to be intra-bursal vs. those patients whose blinded injection was extra-bursal).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Clinical diagnosis of trochanteric bursitis

Exclusion Criteria:

* Pregnancy
* Allergy to contrast
* Untreated coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Numerical pain scores | 1 and 3 month post-injection

SECONDARY OUTCOMES:
SF-36, Oswestry Disability Index, Satisfaction | 1 and 3 months post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Cohen, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Blaustein Pain Treatment Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Cohen SP, Narvaez JC, Lebovits AH, Stojanovic MP. Corticosteroid injections for trochanteric bursitis: is fluoroscopy necessary? A pilot study. Br J Anaesth. 2005 Jan;94(1):100-6. doi: 10.1093/bja/aei012. Epub 2004 Oct 29. PMID 15516348
- [Background] Schapira D, Nahir M, Scharf Y. Trochanteric bursitis: a common clinical problem. Arch Phys Med Rehabil. 1986 Nov;67(11):815-7. PMID 3778178
- [Derived] Cohen SP, Strassels SA, Foster L, Marvel J, Williams K, Crooks M, Gross A, Kurihara C, Nguyen C, Williams N. Comparison of fluoroscopically guided and blind corticosteroid injections for greater trochanteric pain syndrome: multicentre randomised controlled trial. BMJ. 2009 Apr 14;338:b1088. doi: 10.1136/bmj.b1088. PMID 19366755